CLINICAL TRIAL: NCT03816956
Title: A Randomized Double-blind Placebo-controlled Multicenter Phase 3 Study of Efficacy and Safety of AR-301 as Adjunct Therapy to Antibiotics in the Treatment of Ventilator-Associated Pneumonia (VAP) Caused by S. Aureus
Brief Title: Adjunctive Therapy to Antibiotics in the Treatment of S. Aureus Ventilator-Associated Pneumonia With AR-301
Acronym: AR-301-002
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Aridis Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AR-301-002
Record Dates: First submitted 2018-12-21; First posted 2019-01-25 (Actual); Last update posted 2023-07-06 (Actual); Status verified 2023-07

CONDITIONS: Lung Infection; Pneumonia, Ventilator-Associated; Infection, Bacterial; Staphylococcus Aureus
Keywords: Staphylococcus aureus; S. aureus; monoclonal antibody; Aridis; VAP; ventilator acquired pneumonia; infection; pneumonia; AR301
MeSH Terms: conditions — Pneumonia, Ventilator-Associated; Bacterial Infections; Staphylococcal Infections; Infections; Pneumonia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Study treatment (Experimental): Investigational/ Interventional Product group: AR-301 (tosatoxumab) 20 mg/kg administered once intravenously on the day of randomization.
  Interventions: Drug: AR-301
- Placebo treatment (Placebo Comparator): Control group: Placebo administered intravenously on the day of randomization.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: AR-301 — AR-301 (tosatoxumab) 20 mg/kg administered once intravenously the day of enrolment.
  Other Names: AR-301 (tosatoxumab)
  Arms: Study treatment
Other: Placebo — Placebo comparator
  Arms: Placebo treatment

SUMMARY:
AR-301 is being evaluated as an adjunctive treatment of ventilator-associated pneumonia (VAP) due to Staphylococcus aureus (S. aureus) in combination with standard of care (SOC) antibiotic therapy in patients with confirmed S. aureus infection.

DETAILED DESCRIPTION:
This study is an international, multicenter, prospective, randomized, double blind, placebo controlled, parallel design protocol in patients with Ventilator-Associated Pneumonia (VAP) caused by S. aureus.

Patients with a documented diagnosis of pneumonia due to S. aureus, and require ICU care, who have been intubated (or have a tracheostomy tube in place) and mechanically ventilated for at least 48 hours are eligible for screening.

In total, approximately 240 subjects will be randomized 1-1 to be treated with placebo plus standard of care (SOC) or AR-301 (20 mg/kg) plus SOC in this Phase 3 study.

Study subjects will receive a single dose at Day 0 in addition to SOC antibiotic treatment, and then enter a safety, efficacy and PK study period for a total study duration of 28 days. The selection of SOC antibiotics is made in accordance with local best practices at the discretion of the investigator.

ELIGIBILITY:
Inclusion Criteria:

1. Written Informed Consent given by the patient or, if not possible, by a legally acceptable representative and/or an independent physician as authorized by the competent ethics committee (EC) or independent review board (IRB) and local regulations.
2. To be at least 18 years of age. Taiwan only: To be at least 20 years of age. South Korea only: To be at least 19 years of age.
3. Treated in an ICU at the time of enrollment.
4. Endotracheal tube in place (tracheostomy is allowed).
5. The patient is mechanically ventilated for at least 48 hours.
6. Diagnosis of pneumonia based on the following criteria (a, b, and c, all must be met):

   1. One definitive chest X-ray diagnostic of pneumonia within 48 hours,
   2. Hypoxemia based on PaO2/FiO2.
   3. At least one of the following signs:

   i. Documented fever (e.g., body temperature greater than or equal to 38º Celsius).

   ii. Hypothermia (e.g., core body temperature less than or equal to 35º Celsius).

   iii. Total peripheral white blood cell (WBC) count greater than or equal to 10,000 cells/µL (or mm3).

   iv. Leukopenia with total WBC less than or equal to 4,500 cells/µL (mm3). v. Greater than 15 percent immature neutrophils (bands) noted on peripheral blood smear.
7. Documented pulmonary infection with Staphylococcus aureus obtained by bronchoalveolar lavage (BAL), mini-BAL, protected endotracheal aspiration/aspirate (ETA) (collectively 'airway specimen').

Exclusion Criteria

1. The subject is unlikely to survive for the study duration despite delivery of adequate antibiotics and supportive care for treatment of S. aureus pneumonia.
2. Effective antibacterial drug therapy for the index pneumonia administered continuously for 48 hours or more prior to initiation of study treatment. Effective antibiotics would include those typically used to treat S. aureus.
3. Plasmapheresis (ongoing or planned), extracorporeal membrane oxygenation (ECMO) or any procedure that would remove/filter out the monoclonal antibody/study drug.
4. Immunocompromised patients.
5. Known hereditary complement deficiency.
6. Liver dysfunction with a Child Pugh C score > 9 (Child Pugh score of A or B are acceptable at discretion of the Principal Investigator [PI]).
7. Pulmonary disease that precludes evaluation of a therapeutic response (such as lung cancer resulting in bronchial obstruction or on the same side as the pneumonia, active tuberculosis, cystic fibrosis, granulomatous disease, fungal pulmonary infection, lung abscess, pleural empyema or post obstructive pneumonia).
8. Patient has received intravenous (IV) immunoglobulin therapy within 3 months prior to the Screening Visit.
9. Any woman of child-bearing potential (WOCBP) who does not have a negative pregnancy test result at Screening using SERUM or URINE testing based on Beta-subunit human chorionic gonadotropin (HCG) standard tests and methods from the local laboratory.
10. Any sexually active subject who is unwilling to use acceptable methods of contraception for 120 days after dosing.
11. Known lack of treatment compliance from prior studies or ongoing medical care based on medical records and PI's judgment and/or the capacity of the patient to comply with all study requirements.
12. Any medical, psychological, cognitive, social or legal conditions that would interfere in the ability to give an Informed Consent OR the absence of a legally valid representative of the patient or independent physician allowed and able to give consent on his/her behalf.
13. Participation as a subject in another interventional study within 30 days prior to the first dose of study treatment, or planned participation in such a study during the study or within 30 days of its completion by the patient.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 174 (Actual)
Dates: Start 2019-05-03 (Actual); Primary Completion 2022-10-28 (Actual); Study Completion 2022-10-28 (Actual)

PRIMARY OUTCOMES:
A comparison of Clinical Cure Rates of standard of care (SOC) alone and SOC with AR-301 | 21 days
  Clinical cure rates of standard of care (SOC) alone and (SOC) with AR-301 at Day 21 as measured by all-cause mortality, need for mechanical ventilation and signs and symptoms of pneumonia.
Safety of AR-301 by treatment-emergent adverse events assessed by changes between treatment and placebo as assessed by the Principal Investigator | 21 Days
  Safety of AR-301 of treatment-emergent adverse events as assessed by changes assessed by the PI between treatment and placebo
Tolerability of AR-301 measured by the number of participants with treatment-emergent adverse events classified using CTCAE v 5.0 | 21 Days
  Tolerability of AR-301 will be measured and evaluated by the severity of treatment-emergent adverse events using the CTCAE v 5.0.

SECONDARY OUTCOMES:
The difference in clinical cure rates between Standard of Care alone or with AR301 as time to clinical cure at Day 7, 14 and 28 | Day 7, 14, and 28
  Difference in Clinical Cure rates between SOC alone or with AR-301 defined by time to clinical cure (number of days) using the same criteria as for the primary efficacy objective at Day 21.
The difference in mortality between Standard of Care alone or with AR-301 at Days 7,14,28 | Day 7, 14, and 28
  Difference in mortality defined as cause of death (all-cause mortality and pneumonia-related mortality)between SOC alone or with AR-301 at Days 7,14, and 28
The difference in PaO2/FiO2 between Standard of Care alone or with AR-301 at Days 7,14,28 | Day 7, 14, and 28
  Difference in respiratory function between SOC alone or with AR-301 at Days 7,14, and 28 as changes in PaO2/FiO2 ratio (e.g. by arterial blood gases), if available and whenever possible OR changes in non-invasive measures of oxygenation (e.g. by pulse oximetry)
The difference in time on supplemental oxygen assessment between Standard of Care alone or with AR-301 at Days 7,14,28 | Day 7, 14, and 28
  Difference in respiratory function between SOC alone or with AR-301 at Days 7,14, and 28 as time on supplemental oxygen
Changes in baseline in SOFA score between Standard of Care alone or with AR301 at Days 7,14,28 | Day 7, 14, and 28
  Difference in Clinical Cure rates between SOC alone or with AR-301 at Days 7,14, and 28 in the following clinical outcomes:
  Changes from Baseline in sequential organ failure assessment (SOFA) score using the following scale: Maximum SOFA score 0-6, <10% Mortality, 7-9 15-20% mortality, 10-12 40-50% mortality, 13-14 50-60% mortality, 15 >80% mortality, 15-24 >90% mortality. Lower numbers are considered to be better outcome of mortality and higher scores worse outcome of mortality.
Duration of intubation with ventilation | 28 days
  Number of days with intubation with ventilation
Duration mechanical ventilation if tracheostomy in place | 28 days
  Number of days of intubation with mechanical ventilation if tracheostomy in place
Duration of stay in ICU | 28 days
  Number of days of stay in ICU
Duration hospitalization | 28 days
  Number of days of hospitalization
Duration antibiotic use. | 28 days
  Number of days on antibiotics
Pharmacokinetic Analysis - (Cmax) | 28 days
  Pharmacokinetic analysis measuring Maximum Serum Concentration (Cmax)
Pharmacokinetic Analysis - (AUC) | 28 Days
  Pharmacokinetic analysis measuring Area Under the Curve (AUC)
Pharmacokinetic Analysis - (T1/2) | 28 Days
  Pharmacokinetic analysis measuring time for half of the initial dose of study drug to be eliminated from the body (T1/2)
Pharmacokinetic Analysis - (Tmax) | 28 Days
  Pharmacokinetic analysis measuring time at which Cmax is obtained (Tmax)
Pharmacokinetic Analysis (Blood levels of AR-301) | 28 Days
  Blood levels of AR-301 in the patient over time during the study period.

CONTACTS AND LOCATIONS:
Overall Officials: Hasan S Jafri, MD, FAAP, Study Director — Aridis Pharmaceuticals
Locations (45):
- Belarus (3):
  - BLR-06, Grodno
  - BLR-04, Homyel
  - BLR-01, Minsk
- Belgium (2):
  - BEL-01, Lodelinsart
  - BEL-05, Ottignies
- Brazil (2):
  - BRA-08, Curitiba
  - BRA-04, Curitiba
- CHN-09, Guangzhou, Guangdong, China
- EST-01, Tallinn, Estonia
- France (9):
  - FRA-02, Strasbourg, Cedex
  - FRA-18, Brive-la-Gaillarde
  - FRA-10, Bron
  - FRA-05, La Roche-sur-Yon
  - FRA-04, Limoges
  - FRA-01, Nantes
  - FRA-16, Orléans
  - FRA-11, Rennes
  - FRA-13, Trévenans
- Georgia (8):
  - GEO-06, Gori
  - GEO-01, Kutaisi
  - GEO-03, Kutaisi
  - GEO-04, Kutaisi
  - GEO-10, Kutaisi
  - GEO-02, Tbilisi
  - GEO-09, Tbilisi
  - GEO-07, Tbilisi
- Israel (2):
  - ISR-04, Haifa
  - ISR-01, Ramat Gan
- LVA-02, Riga, Latvia
- MEX-07, Guadalajara, Jalisco, Mexico
- Russia (7):
  - RUS-18, Arkhangelsk
  - RUS-11, Chelyabinsk
  - RUS-01, Krasnoyarsk
  - RUS-04, Novosibirsk
  - RUS-02, Saint Petersburg
  - RUS-10, Smolensk
  - RUS-16, Zhukovskiy
- ZAF-09, Johannesburg, South Africa
- ESP-01, Madrid, Spain
- Turkey (Türkiye) (2):
  - TUR-06, Istanbul
  - TUR-01, Trabzon
- Ukraine (4):
  - UKR-05, Chernivtsi
  - UKR-03, Ivano-Frankivsk
  - UKR-02, Kharkiv
  - UKR-09, Kharkiv

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Website of the Sponsor — https://www.aridispharma.com/contact-us/